CLINICAL TRIAL: NCT05893368
Title: New Model for Integrating Person-based Care (PbC) in the Treatment of Advanced HER2-negative Breast Cancer: InPerson Study
Brief Title: New Model for Integrating Person-based Care (PbC) in the Treatment of Advanced HER2-negative Breast Cancer
Acronym: PERGIQUAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID5640
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2023-05

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sharing all key aspects associated with the quality of life in a single digital environment — A digital platform called DNMLAB (DNMLAB) offers the possibility of sharing all key aspects associated with the quality of life in a single digital environment by activating:
  * a digital narrative diary in which the patient has the opportunity to share with the multidisciplinary team her needs, critical issues
  * report Patient-Reported Outcome Measures (PROMs) aimed at detecting health-related quality of life (i.e. QLQ-C30-B23 EORTC).
  * digital narrative diary focused on three main areas of health-related behavior-nutrition, physical activity, and sleep habits-aimed at personalizing and reshaping lifestyle, daily behaviors and, if required, the care pathway.
  The patient will be guided by narrative prompts, but at the same time will always be free to share all aspects related to her lifestyle that she deems useful, in addition to those detected, to benefit from a personalized care approach.

SUMMARY:
The emerging paradigm of person-centered medicine has resulted in a change in the approach and management of health needs, and the introduction of new models and tools into clinical practice. One important change is the introduction of quality of life measurement (HRQoL). The tools used, however, remain anchored in a purely quantitative model, which does not enter the person's specific identity and emotional territory. The perception of quality of life is highly subjective, anchored in each person's needs and expectations (relative deprivation). The structured integration of the patient's point of view can be strengthened by the introduction of narrative medicine and qualitative methodologies, which enrich the point of view expressed in a standardized way, favoring person-centered care and not categories of patients.

The National Chronicity Plan (2016) promotes the application of narrative medicine in clinical practice, aiming at the personalization of care: "the patient-person and his or her individual 'global' health project built through a personalized and shared 'Care Pact' that considers not only his or her clinical condition, but also the life context in which the disease is experienced".

The current spread of digital tools in health care can facilitate the integration of qualitative and quantitative components through the use of dedicated platforms.

In breast cancer patients with advanced disease, especially with triple-negative and HER2-negative biological subtype, oncological treatments include chemotherapy regimens, without or with target therapies and biological treatments combined with endocrinotherapy. For these patients, there is a need to improve treatment-related outcomes and overall quality of care and quality of life. To date, there is a lack of detection of subjective experience on an ongoing basis, which is the basis for personalization of care, and which may also have an impact on adherence to cancer treatment.

The study aims to evaluate the introduction of the digital Person based Care (PbC) model designed by the project team. The model uses an online platform to integrate HRQoL quantitative data and qualitative narrative data for personalized care pathway based on the daily needs and existential project of the patient/caregiver.

DETAILED DESCRIPTION:
The healthcare system has undergone significant changes with the emergence of a person-centered medicine paradigm. Nowadays, care pathways are evaluated not only based on clinical results, but also on their impact on patients' quality of life. With the medical and therapeutic advancements in healthcare, the need for more integrated, empathic, and person-centered clinical approaches that consider the needs and expectations of patients is growing.

Clinical practice has introduced new measurement tools to capture the patient's perspective on the outcomes of care pathways, including Patient-Reported Outcome Measures (PROMs) aimed at evaluating patients' perceived quality of life during treatment and follow-up. However, currently approved questionnaires do not exhaustively inform clinicians on how disease and treatments impact a patient's care journey.

In this context, narrative medicine has proven to be a valid and reliable methodology for integrating the patients' perspective into standard clinical evaluation. Qualitative methodologies provided by narrative medicine can enrich the information expressed in standardized questionnaires, allowing access to the existential and emotional components of the patients' care experience. Narrative medicine can capture the perception of quality of life, which is highly subjective and influenced by each individual's needs and expectations (i.e. relative deprivation).

Systematic collection of patient-reported outcomes (PROs) has proven to be a valid, reliable, and accurate methodology in oncology for assessing care pathway outcomes and monitoring drug toxicity, as impacts and symptoms may be overlooked or underestimated by the clinicians. Narrative medicine has also proven to be feasible and reliable in improving physician-patient communication and promoting a bio-psycho-social personalization of the care pathway, particularly when used with digital listening tools, such as the digital narrative diary. Studies on digital narrative medicine in oncology have shown the potential of digital platforms in promoting the listening of patients' needs by a multidisciplinary team throughout the care pathway, resulting in a positive impact not only on the patient but also on the healthcare team.

The transition from a traditional disease-centered to a more person-centered care model has led to the introduction of integrative medicine in oncological care centers. Through a rational and evidence-based use of lifestyles, psychological support and complementary therapies, integrative medicine promotes better control of side effects, greater adherence to treatment protocols, and optimization of the patients' quality of life throughout their care pathway. In the context of breast, integrative oncology combines conventional oncological treatments with integrative therapies to support individuals in their bio-psycho-social dimension, thus providing effective and minimally invasive responses to complex and sometimes unmet health needs.

The objective of this project is to employ these resources in a digital listening and communication pathway to benefit the quality of life of patients affected by HER2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient able to understand, sign and date the informed consent prior to any specific study procedure;
* Diagnosis of HER2-negative advanced breast cancer (ER and PgR hormone receptor negative or ER and/or PgR receptor positive), undergoing cancer treatment
* Age ≥18 years
* Knowledge of the Italian language
* Life expectancy ≥ 24 weeks
* Basic level of digital knowledge.

Exclusion Criteria:

* Inability to participate in the patient's study (psychiatric disorders, PS ECOG > 2) and unavailability of caregiver;
* Unavailability of an e-mail account or unavailability to use web-based tools (for the patient/caregiver);
* Patients who do not sign informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with HER2-negative advanced breast cancer (IHC score 0, 1+, or 2+ with non-amplified FISH/SISH) on 1st or 2nd line treatment, with advanced disease, under oncological treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Standardized quality of life measurement | 12 months
  ● The integration of standardized quality of life measurement with the patient's subjective narrative through the application of validated narrative medicine methodologies.
Perceived quality of life | 12 months
  The improvement of perceived quality of life for patients with advanced breast cancer.
Personalization of care pathway | 12 months
  The personalization of the care pathway with integrative therapies, based on the patients' needs, attitudes and lifestyles.
Improvement of quality of life | 12 months
  The improvement of the quality of the patient-physician relationship.

SECONDARY OUTCOMES:
Validation of digital tools | 12 months
  The validation of digital tools to introduce innovative models of patient engagement and compliance in the care pathway.
Enhancement of communicative processes | 12 months
  The enhancement of communicative processes aimed at informing metastatic patients about the most suitable lifestyles to positively impact their quality of life.
Patients' awareness regarding their own disease condition | 12 months
  The increase of patients' awareness regarding their own disease condition, treatment effects, and care needs that may arise during treatment.
Strengthening of multidisciplinary team | 12 months
  The strengthening of the multidisciplinary team interaction
Enhancement of information exchange and sharing of experiences among patients with the same condition | 12 months
  The enhancement of information exchange and sharing of experiences among patients with the same condition in a privacy-protected digital environment.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico A. Gemelli - IRCCS, Rome, Italy

REFERENCES:
- [Derived] Fabi A, Rossi A, Mocini E, Cardinali L, Bonavolonta V, Cenci C, Magno S, Barberi V, Moretti A, Besharat ZM, Iolascon G, Baldari C, Ferretti E, Botticelli A, Paris I, Scambia G, Migliaccio S. An Integrated Care Approach to Improve Well-Being in Breast Cancer Patients. Curr Oncol Rep. 2024 Apr;26(4):346-358. doi: 10.1007/s11912-024-01500-1. Epub 2024 Feb 24. PMID 38400984